CLINICAL TRIAL: NCT07016893
Title: Exercise Workshop, Skill-Based Art Approaches, and Awareness Studies for Elderly Individuals With Cognitive Impairment
Brief Title: Exercise Workshop, Skill-Based Art Approaches, and Awareness Studies for Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Pamukkale University (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gulfidan Tokgoz, Balıkesir University, Balikesir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024/112
Record Dates: First submitted 2025-06-03; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia; Alzheimer Disease; Geriatric Rehabilitation; Elderly (People Aged 65 or More)
Keywords: Mild Cognitive Impairment; dementia; alzheimer's disease; awareness; workshop; art; exercise; elderly health
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise, art, awareness group (Experimental): Mild cognitive impairment (MCI) is an important risk factor for Alzheimer's disease (AD) (Hwang and Lee, 2017). The literature emphasizes that the prevalence of MCI and AD will continue to increase and draws attention to this area (Realdon et al., 2016). The MCI stage, which is the most active part of AD, provides a "window of opportunity" for the prevention and treatment of AD (Wu, 2020). Early prevention strategies are considered important, especially during this period. Improving the individual's cognitive functions and reducing symptoms in the MCI stage will reduce the incidence of AD, thereby reducing healthcare costs and improving the individual's condition and quality of life (Jak, 2012). Since AD is irreversible and faces significant treatment challenges, the key to preventing and treating the disease is to take early prevention and intervention measures (Zhang et al., 2021). When considering these interventions, focus is placed on potentially modifiable risk factors that ma
  Interventions: Other: Healthy aging interventions

INTERVENTIONS:
Other: Healthy aging interventions — In our study workshop activities conducted for eight weeks and included an Exercise Workshop (Music-Based Exercise Workshop, Exercise Training with Active Video Games (Exergaming), Clinical Pilates Training Workshop, Cognitive Exercise Therapy Approach Workshop, Nordic walking, dance therapy), Skill-Oriented Art Workshop (Systemic Calligraphy Therapy Workshop, soap-candle making workshop, culinary arts workshop), and Disease Awareness Studies (disease awareness information and education, the process from diagnosis to acceptance, experiences of patients and relatives, use of daily life technologies, home adjustments against falls, introduction of municipal services for the elderly).

SUMMARY:
Purpose: The aim of the project is to contribute to the physical, social, and psychological well-being of elderly individuals with cognitive impairment within a multidisciplinary approach framework, and to increase the level of knowledge and awareness about diseases and aging by organizing exercise, art, and education workshops under the guidance of expert health and art professionals.

Scope and Target Group: Cognitive impairment affects daily life activities by impacting cognitive abilities such as memory, attention, and concentration. Mild Cognitive Impairment (MCI), Dementia, and Alzheimer's Disease (AD) are common cognitive impairments in the elderly. Early prevention strategies and intervention measures during this period are crucial. It is known that non-pharmacological interventions, especially in the early stages of MCI, are a window of opportunity that is promising and cost-effective. The primary target audience of this project is elderly individuals diagnosed with MCI, Dementia, and AD. To maximize the impact, some of the planned training sessions included family members of patients.

Method and Expected Results: The project carried out in collaboration with Balıkesir University and Balıkesir Altıeylül Municipality. Various exercise and art workshops organized. Workshop activities conducted for eight weeks and included an Exercise Workshop (music-based exercises, exercise with active video games, clinical Pilates training, cognitive exercise therapy approach, Nordic walking, dance therapy), Skill-Oriented Art Workshop (systemic calligraphy therapy, soap-candle making workshop, culinary arts workshop), and Disease Awareness Studies (disease awareness information and education, the process from diagnosis to acceptance, experiences of patients and relatives, use of daily life technologies, home adjustments against falls, introduction of municipal services for the elderly).

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years of age
* Having one of the diagnoses of MCI, dementia, or Alzheimer's by a neurologist or geriatrician
* Having less than 27 points on the Mini Mental State Examination (Zhuang et al., 2021).
* Being between stages 2-5 on the Global Impairment Scale.

Exclusion Criteria:

* Having a pulmonary, neurological, musculoskeletal, or rheumatological disease that may prevent exercise
* Having balance problems or lower extremity asymmetry at a level that may prevent exercise
* Individuals with unstable medical conditions (uncontrolled diabetes or hypertension, deep vein thrombosis, etc.)
* Having vision or hearing problems at a level that will prevent participation in workshops

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-09-28 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Test | From enrollment to the end of intervention at 8 weeks
  It is emphasized in the literature that the Mini Mental State Examination (MMST) is the most frequently used test worldwide for cognitive disorders (Ciesielska et al., 2016). MMST tests orientation, memory, attention, calculation, recall, language, motor function and perception, and visuospatial abilities, and its greatest advantage is that it can be applied easily and quickly (Salis et al., 2023). MMST was used to evaluate cognitive functions in our study. A score between 27-30 on the MMST is considered normal, 24-27 as MCI, 20-23 as mild stage, 10-19 as moderate stage, and 0-9 as advanced stage dementia (Güngen et al., 2002). Individuals with a score of 27 or less on the MMST were included in our study.
Montreal Cognitive Assessment Scale (MoCA) | From enrollment to the end of intervention at 8 weeks
  MoCA is one of the most frequently used tools in clinics to assess cognitive functions and has been translated into 35 languages (Sokolowska et al., 2018). It tests many cognitive domains including short-term memory, visual-spatial skills, executive functions, attention, concentration and working memory, language and orientation. It has been reported that its sensitivity varies between 67-100% and its specificity between 50-95% when evaluated using different cutoffs (Zhuang et al., 2021). The advantage of the test is that it provides a more comprehensive assessment compared to the assessment methods used in the field and is used quite frequently in the elderly population (Breton et al., 2019). MoCA was used in the project to assess the change in cognitive functions of individuals with cognitive impairment.

SECONDARY OUTCOMES:
Muscle Strength Assessment | From enrollment to the end of intervention at 8 weeks
  Handgrip strength is a suitable measurement method for both clinical practice and public health research. Although the measurement of handgrip strength evaluates the function of a muscle group, it can be used to obtain a general idea about the musculoskeletal system in older adults. For this reason, it has been accepted as an indicator of general body strength. In our study, hand dynamometer and pinchmeter devices were used to evaluate the muscle strength of the participants. For the measurement of handgrip strength, participants were asked to sit in a chair with back support and fixed arms and rest their forearms on the arm of the chair so that their wrists were just at the edge of the chair. Measurements were made three times with a hand dynamometer, one minute apart, from the right and left hands, and the average of the results was recorded (Vermeulen et al., 2015).
Flexibility Assessment | From enrollment to the end of intervention at 8 weeks
  Spinal mobility and flexibility are an important component of healthy physical fitness for elderly individuals (Taşpınar et al., 2023). One of the methods frequently used in the literature for flexibility assessment is the sit-and-reach test. The patient is asked to sit with their legs together and their feet on a box, then bend forward as much as possible by extending their arms, without bending their knees, and remaining motionless for 1-2 seconds. The measurement was repeated three times and the average of the farthest distances reached was recorded in cm (Mayorga-Vega et al., 2014).
Physical Activity Level | From enrollment to the end of intervention at 8 weeks
  The short form of the International Physical Activity Questionnaire (IFQQ) was used to determine the physical activity levels of the participants. The IFQQ is a 7-item scale that evaluates the duration and frequency of vigorous physical activity, moderate physical activity, walking and sedentary behavior based on MET values (Craig et al., 2003). The physical activity levels were calculated according to the scores obtained by multiplying the duration, frequency and MET values of the physical activities that the participants participated in for at least 10 minutes within 7 days. The physical activity level assessment was made at the beginning and end of the project, and was repeated three months after the workshops were completed to evaluate sustainability.
Depression Assessment | From enrollment to the end of intervention at 8 weeks
  The Elderly Depression Scale (GDS) is a tool for the diagnosis and assessment of depression in elderly individuals and was developed based on the findings that elderly individuals with depression exhibit unique symptoms such as physical symptoms, anxiety, and decreased cognitive functions (Sheline et al., 2006).
Quality of Life Assessment | From enrollment to the end of intervention at 8 weeks"
  Quality of life is a concept related to the individual's perception of his/her situation in life in line with his/her expectations, goals, interests and desires within the culture and social environment he/she lives in, and is defined as the multidimensional evaluation of the individual's person-environment system according to both personal and socio-economic criteria (Stoner et al., 2019). In our study, the 19-item Quality of Life Scale for the Elderly, developed by Hyde et al. (2003), specific to the elderly population, was used.
Well-Being of Individuals Who Provide Care | From enrollment to the end of intervention at 8 weeks
  Caregiving, which is a multidimensional experience, can cause difficulties as well as positive aspects. In our study, the "Zarit Caregiving Burden Scale" was used to assess the stress experienced by those who provide care to elderly individuals. Studies have reported that the internal consistency coefficient of the scale is between 0.87-0.94 and the test-retest reliability is 0.71. The scale, which can be filled out by the caregivers themselves or the researcher, consists of 22 items that determine the effect of caregiving on the individual's life. The Likert-type scale can also be answered as never, rarely, sometimes, often, or almost always. The minimum score that can be obtained from the scale is 0 and the maximum score is 88. A high scale score indicates that the distress experienced is high.
Satisfaction, Knowledge and Awareness Assessment | From enrollment to the end of intervention at 8 weeks
  At the end of all workshops, patient and caregiver satisfaction, exercise or disease-related knowledge and awareness levels were evaluated by the research team according to the content of the activity. Patients and their relatives were asked to rate their satisfaction level out of 10 after the activities and to answer questions about satisfaction. Below are sample questions that we want the patient to rate as strongly agree (5), agree (4), undecided (3), disagree (2), strongly disagree (1):
  * I had a good time and enjoyed the workshop.
  * The training of expert staff increased my awareness of methods for combating the disease.
  * Workshops increased my social participation.
  * I am aware that I need to gain an exercise habit in order to increase my physical activity level.
  * Exercise, art and music increase my quality of life and psychological well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University Cagis Campus 10145 Balikesir, Balıkesir, Balikesir University Cagis Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoner CR, Orrell M, Spector A. The psychometric properties of the control, autonomy, self-realisation and pleasure scale (CASP-19) for older adults with dementia. Aging Ment Health. 2019 May;23(5):643-649. doi: 10.1080/13607863.2018.1428940. Epub 2018 Jan 22. PMID 29356567
- [Background] Shin C, Park MH, Lee SH, Ko YH, Kim YK, Han KM, Jeong HG, Han C. Usefulness of the 15-item geriatric depression scale (GDS-15) for classifying minor and major depressive disorders among community-dwelling elders. J Affect Disord. 2019 Dec 1;259:370-375. doi: 10.1016/j.jad.2019.08.053. Epub 2019 Aug 20. PMID 31470180
- [Background] Sheline YI, Barch DM, Garcia K, Gersing K, Pieper C, Welsh-Bohmer K, Steffens DC, Doraiswamy PM. Cognitive function in late life depression: relationships to depression severity, cerebrovascular risk factors and processing speed. Biol Psychiatry. 2006 Jul 1;60(1):58-65. doi: 10.1016/j.biopsych.2005.09.019. Epub 2006 Jan 18. PMID 16414031
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Mayorga-Vega D, Merino-Marban R, Viciana J. Criterion-Related Validity of Sit-and-Reach Tests for Estimating Hamstring and Lumbar Extensibility: a Meta-Analysis. J Sports Sci Med. 2014 Jan 20;13(1):1-14. eCollection 2014 Jan. PMID 24570599
- [Background] Taspinar G, Angin E, Oksuz S. The effects of Pilates on pain, functionality, quality of life, flexibility and endurance in lumbar disc herniation. J Comp Eff Res. 2023 Jan;12(1):e220144. doi: 10.2217/cer-2022-0144. Epub 2022 Dec 1. PMID 36453667
- [Background] Vermeulen J, Neyens JC, Spreeuwenberg MD, van Rossum E, Hewson DJ, de Witte LP. Measuring grip strength in older adults: comparing the grip-ball with the Jamar dynamometer. J Geriatr Phys Ther. 2015 Jul-Sep;38(3):148-53. doi: 10.1519/JPT.0000000000000034. PMID 25594521
- [Background] Breton A, Casey D, Arnaoutoglou NA. Cognitive tests for the detection of mild cognitive impairment (MCI), the prodromal stage of dementia: Meta-analysis of diagnostic accuracy studies. Int J Geriatr Psychiatry. 2019 Feb;34(2):233-242. doi: 10.1002/gps.5016. Epub 2018 Nov 27. PMID 30370616
- [Background] Zhuang L, Yang Y, Gao J. Cognitive assessment tools for mild cognitive impairment screening. J Neurol. 2021 May;268(5):1615-1622. doi: 10.1007/s00415-019-09506-7. Epub 2019 Aug 14. PMID 31414193
- [Background] Sokolowska N, Sokolowski R, Polak-Szabela A, Mazur E, Podhorecka M, Kedziora-Kornatowska K. Comparison of the effectiveness of the Montreal Cognitive Assessment 7.2 and the Mini-Mental State Examination in the detection of mild neurocognitive disorder in people over 60 years of age. Preliminary study. Psychiatr Pol. 2018 Oct 27;52(5):843-857. doi: 10.12740/PP/68611. Epub 2018 Oct 27. English, Polish. PMID 30584818
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Salis F, Costaggiu D, Mandas A. Mini-Mental State Examination: Optimal Cut-Off Levels for Mild and Severe Cognitive Impairment. Geriatrics (Basel). 2023 Jan 12;8(1):12. doi: 10.3390/geriatrics8010012. PMID 36648917
- [Background] Ciesielska N, Sokolowski R, Mazur E, Podhorecka M, Polak-Szabela A, Kedziora-Kornatowska K. Is the Montreal Cognitive Assessment (MoCA) test better suited than the Mini-Mental State Examination (MMSE) in mild cognitive impairment (MCI) detection among people aged over 60? Meta-analysis. Psychiatr Pol. 2016 Oct 31;50(5):1039-1052. doi: 10.12740/PP/45368. English, Polish. PMID 27992895
- [Background] Zhang XX, Tian Y, Wang ZT, Ma YH, Tan L, Yu JT. The Epidemiology of Alzheimer's Disease Modifiable Risk Factors and Prevention. J Prev Alzheimers Dis. 2021;8(3):313-321. doi: 10.14283/jpad.2021.15. PMID 34101789
- [Background] Jak AJ. The impact of physical and mental activity on cognitive aging. Curr Top Behav Neurosci. 2012;10:273-91. doi: 10.1007/7854_2011_141. PMID 21818703
- [Background] Wu C, Yang L, Li Y, Dong Y, Yang B, Tucker LD, Zong X, Zhang Q. Effects of Exercise Training on Anxious-Depressive-like Behavior in Alzheimer Rat. Med Sci Sports Exerc. 2020 Jul;52(7):1456-1469. doi: 10.1249/MSS.0000000000002294. PMID 32028456
- [Background] Realdon O, Rossetto F, Nalin M, Baroni I, Cabinio M, Fioravanti R, Saibene FL, Alberoni M, Mantovani F, Romano M, Nemni R, Baglio F. Technology-enhanced multi-domain at home continuum of care program with respect to usual care for people with cognitive impairment: the Ability-TelerehABILITation study protocol for a randomized controlled trial. BMC Psychiatry. 2016 Nov 25;16(1):425. doi: 10.1186/s12888-016-1132-y. PMID 27887597
- [Background] Hwang J, Lee S. The effect of virtual reality program on the cognitive function and balance of the people with mild cognitive impairment. J Phys Ther Sci. 2017 Aug;29(8):1283-1286. doi: 10.1589/jpts.29.1283. Epub 2017 Aug 10. PMID 28878448
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27887597/